CLINICAL TRIAL: NCT00533520
Title: Evaluation of Dosing Interval of Higher Doses of Ranibizumab
Acronym: BGB/IST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brandon G. Busbee, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Brandon G. Busbee, MD, Sponsor-Investigator, Tennessee Retina
Organization: Tennessee Retina (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4155s
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.5mg ranibizumab (Active Comparator): Subjects will be treated with 0.5mg ranibizumab at the Day 0 visit and the as needed based on defined retreatment criteria no sooner than every 28 days since last treatment.
  Interventions: Drug: ranibizumab
- 1.0mg ranibizumab (Active Comparator): Subjects will be treated with 1.0mg ranibizumab at the Day 0 visit and the as needed based on defined retreatment criteria no sooner than every 28 days since last treatment.
  Interventions: Drug: ranibizumab
- 2.0mg ranibizumab (Active Comparator): Subjects will be treated with 2.0 mg ranibizumab at the Day 0 visit and the as needed based on defined retreatment criteria no sooner than every 28 days since last treatment.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Arm A: 0.5 mg ranibizumab on day 0 with retreatment based on defined criteria not to occur sooner than every 28 days Arm B: 1.0 mg ranibizumab on day 0 with retreatment based on defined criteria not to occur sooner than every 28 days Third Arm 2.0mg Arm with retreatment based on defined criteria not to occur sooner than every 28 days
  Other Names: rhuFab V2

SUMMARY:
Evaluation of Dosing Interval of Higher Doses of Ranibizumab for patients with wet age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Phase 4 study to test the safety, tolerability and effectiveness of a higher doses (1.0 mg and 2.0 mg) of ranibizumab versus the standard dose (0.5 mg), in adults with age related macular degeneration who have never been treated with ranibizumab. An additional purpose is to determine if the higher doses (1.0 mg and 2.0 mg) of ranibizumab can increase the time between doses beyond that currently needed with the 0.5 mg dose.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive macular degeneration patients with choroidal neovascularization
* >50 years old
* Visual acuity 20/40 to 20/320

Exclusion Criteria:

* Pregnancy
* Previous history of thromboembolic event including myocardial infarction or stroke

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety - Presence of intraocular inflammation following intravitreal ranibizumab injection | 24 months

SECONDARY OUTCOMES:
Injection interval: mean time and number of injections | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G Busbee, MD, Principal Investigator — Tennessee Retina, P.C,.
Locations (1):
- Tennessee Retina, P.C., Nashville, Tennessee, United States